CLINICAL TRIAL: NCT01519778
Title: Phase 2 Open-Label Safety and Exploratory Skin Lesion Measurement Study of 6-Day Oral TR-701 FA in Skin Abscess and Cellulitis Patients
Brief Title: A Phase 2 Safety and Exploratory Skin Lesion Measurement of TR-701 FA Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1986-011; TR701-126 (Other: TriusRX Unique ID)
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Major Cutaneous Abscess; Cellulitis; Erysipelas
MeSH Terms: conditions — Cellulitis; Erysipelas | interventions — tedizolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TR-701 FA (Experimental)
  Interventions: Drug: TR701 FA

INTERVENTIONS:
Drug: TR701 FA — 1 tablet 200 mg once daily
  Other Names: Tedizolid

SUMMARY:
Characterization of the safety profile of TR-701 Free Acid (FA) in patients with major cutaneous abscess or cellulitis/erysipelas.

DETAILED DESCRIPTION:
This is an open-label, multicenter study of oral TR-701 FA 200 mg once daily for 6 days for the treatment of major cutaneous abscess or cellulitis/erysipelas in patients 18 years of age or older. This study is designed to further characterize the safety profile and gather additional lesion measurement data of TR-701 FA in patients with major cutaneous abscess or cellulitis/erysipelas.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Suspected or documented gram-positive infection from baseline Gram stain or culture.
* Cellulitis/erysipelas or major cutaneous abscesses at Screening

Exclusion Criteria:

* Postsurgical or open wound infections
* Severe sepsis or septic shock
* Uncomplicated skin and skin structure infections such as furuncles, minor abscesses (< 75 cm2 or area of suppuration not surrounded by cellulitis/erythema), and impetiginous lesions
* Infections associated with, or in close proximity to, a prosthetic device
* Known bacteremia or osteomyelitis at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2012-08-27 (Actual); Study Completion 2012-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (10):
- United States (10):
  - Trius Investigator Site #118, Anaheim, California
  - Trius Investigator Site #129, Buena Park, California
  - Trius Investigator Site 103, Chula Vista, California
  - Trius Investigator Site 105, La Mesa, California
  - Trius Investigator Site #106, Long Beach, California
  - Trius Investigator Site 104, Oceanside, California
  - Trius Investigator Site 101, Columbus, Georgia
  - Trius Investigator Site 102, Savannah, Georgia
  - Trius Investigator Site 128, Las Vegas, Nevada
  - Trius Investigator Site 115, Somers Point, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Powers JH 3rd, Das AF, De Anda C, Prokocimer P. Clinician-reported lesion measurements in skin infection trials: Definitions, reliability, and association with patient-reported pain. Contemp Clin Trials. 2016 Sep;50:265-72. doi: 10.1016/j.cct.2016.08.010. Epub 2016 Aug 13. PMID 27530088

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TR-701 FA
Started | 200
Completed | 186
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | TR-701 FA
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 129

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety will be assessed through summaries of the incidence of AEs and SAEs as well as through summaries of vital signs, physical examinations, ECG findings, and laboratory assessments (hematology, serum chemistry, and urinalysis).
Time Frame: 24-31 days
Population: Patients receiving any amount of study drug
Measure: Number; unit: participants
Arm/Group | TR-701 FA
Number analyzed (Participants) | 200
participants | 91

ADVERSE EVENTS:
Time Frame: From the Informed Consent Form signature through the late follow-up visit, up to 32 days.
Arm/Group | TR-701 FA
Serious Adverse Events (participants affected / at risk) | 2/200
Other Adverse Events (participants affected / at risk) | 58/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TR-701 FA (N=200)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
thrombophlebitis septic (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TR-701 FA (N=200)
Nausea (Gastrointestinal disorders) | 22
diarrhea (Gastrointestinal disorders) | 13
cellulitis (Infections and infestations) | 10
abscess (Infections and infestations) | 9
vomiting (Gastrointestinal disorders) | 9
dizziness (Nervous system disorders) | 7
headache (Nervous system disorders) | 7
chills (General disorders) | 4
constipation (Gastrointestinal disorders) | 4
somnolence (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trius intends to pursue publication of the results of the study in cooperation with a lead Investigator, subject to the terms and conditions of the clinical study agreement between Trius and Investigators. Trius written approval is required for publication of any data subsets. Final authorship will be determined in accordance with the International Conference of Medical Journal Editors definition of authorship.